CLINICAL TRIAL: NCT01918696
Title: Controlled Evaluation of a Computerized Anger-reduction Treatment for Suicide Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jesse Cougle, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013.10885
Record Dates: First submitted 2013-07-11; First posted 2013-08-08 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Anger; Suicidal Ideation
Keywords: suicide; anger; interpretation modification; computerized treatment
MeSH Terms: conditions — Suicidal Ideation; Suicide | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Anger Reduction Treatment (Experimental): This treatment consists of eight 15-minute sessions. Participants will read scenarios and imagine themselves in these situations: "A driver does not let you over even though you have your blinker on." Next, another will appear to provide a less ambiguous interpretation. One letter will be missing from the key word of this sentence. The sentence will read "They can't s_e you." The participant will fill in the missing letter (to form "see"). Next, this interpretation will be reinforced by requiring the participants to correctly answer "yes" or "no" to a comprehension question ("Is the driver being disrespectful?"). In each session 64 training scenarios will be presented. Participants will never see the same scenario twice over the course of the study.
  Interventions: Behavioral: Anger Reduction Treatment
- Progressive Muscle Relaxation (Active Comparator): Participants will receive eight 15-minute sessions of PMR. They will listen to a PMR script (Kassinove & Tafrate, 2002). Participants will be asked to make sure they are sitting comfortably, close their eyes, and systematically tense and release 10 different muscle groups. At the end of this procedure, participants will create a plan for when they will use the exercise. They will then type out the sentence: "When I feel [write the feeling you decided on], then I will use this relaxation technique." They will then be told, "Now, go over what you have written and say it quietly to yourself until you can repeat it word for word without having to read what you have written."
  Interventions: Behavioral: Progressive Muscle Relaxation
- Control Condition (Placebo Comparator): To control for expectancy effects, participants assigned to the control condition will complete eight computerized sessions consisting of psychoeducation on healthy behaviors. These sessions will be matched for time with the active conditions, lasting 15 minutes each. Psychoeducation will cover the topics of exercise, diet, hygiene, social support, healthy activities, and sleep, and will be taken from protocols developed from our ongoing research. This psychoeducation is perceived as credible but has no detectable impact on behavior. After the post-treatment session, participants will be provided with the active ART treatment free of charge if they wish to receive it.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Anger Reduction Treatment — Eight 15-minute sessions of interpretation modification to reduce angry interpretation biases.
  Arms: Anger Reduction Treatment
Behavioral: Progressive Muscle Relaxation — Eight 15-minute sessions of progressive muscle relaxation (PMR) including formulation of a plan to use PMR when angry.
  Arms: Progressive Muscle Relaxation
Behavioral: Control Condition — Eight 15-minute sessions of informative videos on healthy living.
  Arms: Control Condition

SUMMARY:
The purpose of this study is to determine whether a computerized intervention designed to reduce anger-provoking interpretation biases will reduce suicide risk among individuals with elevated levels of trait anger.

DETAILED DESCRIPTION:
Problematic anger is often found among returning military veterans, especially those exposed to combat. Anger control problems are associated with difficulties with reintegration. One study of Iraq-Afghanistan combat veterans who used VA medical services (N = 754) found that difficulty controlling anger was the most commonly reported problem experienced since homecoming, occurring among 57% of the sample (Sayer et al., 2010). Problematic anger and hostility have also been linked to risk for suicide (Daniel et al., 2009; Lehnert, Overholser, & Spirito, 1994; Maiuro, O'Sullivan, Michael, & Vitaliano, 1989). From the perspective of the interpersonal-psychological theory of suicide (Joiner, 2005), individuals with problematic anger may be at increased risk for suicide because they engage in impulsive behaviors (e.g., aggression, substance abuse) intended to manage anger. Such behaviors may lead to exposure to painful and provocative events, which increase their acquired capability for engaging in suicidal behavior. Additionally, anger problems often lead to social isolation, which may contribute to greater perceived burdensomeness and a failed sense of belonging, established risk factors for suicide (Van Orden et al., 2010).

Anger prone individuals are likely to hold the hostile attribution bias, which reflects the tendency to interpret the ambiguous actions of others as reflecting hostile intent (Wilkowski & Robinson, 2008). Recently, researchers have developed computerized interpretation bias modification (IBM) protocols intended to efficiently reduce interpretive biases. These treatments have shown efficacy in reducing anxiety and depression (Beard & Amir, 2008; Holmes, Lang, & Shah, 2009; Mathews et al., 2007). We have conducted studies using similar procedures that focus on hostile interpretation biases and found our program to successfully reduce anger and hostility.

To evaluate the efficacy of the IBM protocol we have developed in reducing anger and suicide risk, we will conduct a three-arm randomized controlled trial over the internet. Military veterans and non-veteran community participants reporting elevated trait anger (N = 120) will be randomized to one of three conditions: 1) IBM; 2) progressive muscle relaxation (PMR); or 3) healthy education videos (control). Each condition will consist of eight 15-minute treatment sessions. Participants will complete two sessions per week for four weeks and will be administered assessments at pre- and post-treatment. IBM and PMR conditions will also complete 3-month and 6-month follow-up assessments. To ensure an adequate test of the effects of this intervention on suicide risk, we will oversample for individuals with current suicidal ideation. We hypothesize that: 1) IBM will lead to greater reductions in anger than PMR and control conditions in a sample with problematic anger; 2) IBM will lead to greater reductions in suicidal ideation, perceived burdensomeness, and thwarted belongingness than PMR and control conditions; 3) efficacy of the IBM condition in reducing suicidal ideation will be mediated by reductions in perceived burdensomeness and thwarted belongingness; 4) group differences between IBM and PMR will be maintained at the 3-month and 6-month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* elevated levels of trait anger (scoring 19 or higher, or the top 25% of the general population)
* must have access to a computer with an internet connection
* must also be English speakers

Exclusion Criteria:

* currently receiving therapy for problematic anger
* evidence of serious suicidal intent requiring hospitalization or immediate treatment
* evidence of psychotic-spectrum disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
State-Trait Anger Expression Inventory-2 (STAXI-2; Spielberger, 1999) | change from baseline at 1-month, 3-months, and 6-months

SECONDARY OUTCOMES:
Beck Suicide Scale (BSS; Beck et al., 1979) | change from baseline at 1-month, 3-months, and 6-months

OTHER OUTCOMES:
Interpersonal Needs Questionnaire (INQ; Van Orden, Cukrowicz, Witte, & Joiner, 2012 | change from baseline at 1-month, 3-month, and 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Jesse R Cougle, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Department of Psychology, Tallahassee, Florida, United States